CLINICAL TRIAL: NCT03420989
Title: Development of a Novel Healthy Snacks Including Seaweeds and Carob Which Improve Risk Factors Associated With Metabolic Syndrome
Brief Title: Elaboration of New Generation Snacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endocrinology and Clinical Nutrition Research Center, Spain (Other)
Responsible Party: Principal Investigator, Daniel de Luis Roman, Medical Doctor, Endocrinology and Clinical Nutrition Research Center, Spain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: casve-nm-15-220
Record Dates: First submitted 2016-12-17; First posted 2018-02-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Snack Food
Keywords: carob; seaweed; snack food; obese subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active snack food (Active Comparator): snack food with carob and seaweeds 50 gr per day
  Interventions: Other: Active snack food
- Control snack food (Placebo Comparator): snack food without carob and seaweeds 50 gr per day
  Interventions: Other: Control snack food

INTERVENTIONS:
Other: Active snack food — snack enriched with seaweeds and carob
  Arms: Active snack food
Other: Control snack food — the same snack food without seaweeds and carob
  Arms: Control snack food

SUMMARY:
It is a blind randomized clinical trial of nutritional intervention in humans with a snack (seaweeds and carob), compared to a control snack without the bioactive ingredients studied but of similar nutritional composition, to evaluate the effect on the lipid profile, glycemia and Insulin resistance.

DETAILED DESCRIPTION:
The design will consist of a double-blind randomized study in adult subjects with metabolic syndrome, who will consume snack (enriched in seaweeds and carob) (50 g / day) vs. conventional snack for 8 weeks.

All the next parameters will be measured/calculated at basal time and after 8 weeks of intervention. The next biochemical parameters will be measured: Total cholesterol, LDL cholesterol, HDL, triglycerides will be analyzed using an enzyme-colorimetric method (Roche Diagnostics , Mannheim, Germany). Glucose will be determined by the method of glucose oxidase (Glucose analyzer 2, Beckman Instruments, Fullerton, California), insulin will be determined by Elisa (ELISA Diagnostic Corporation, Los Angeles, CA) and HOMA will be calculated by the formula Matthew et al. , 1985 (HOMA = (glucose * insulin) / 22.5). Body weight and fat mass by bioimpedance will be measured, too. Blood pressure (Systolic and diastolic blood pressure) will be measured, too. A diet records for 3 days and a satiety scale will be performed at the beginning and end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* presence of metabolic syndrome by (Adult Treatment Panel III) criteria

Exclusion Criteria:

* consume supplements (vitamins, minerals or other dietary components),
* non-restrictive diet
* known chronic disease (eg diabetes, cardiovascular disease, Inflammatory diseases).
* active cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Lipoproteins | change from baseline HDL cholesterol (mg/dl) and LDL cholesterol (mg/dl )levels at 8 weeks
  change in serum lipoprotein levels such as HDL-cholesterol and LDL cholesterol (mg/dl)

SECONDARY OUTCOMES:
carbohydrate metabolism | change from baseline fasting glucose levels (mg/dl) at 8 weeks
  change of seric carbohydrate parameters markers such as fasting glucose levels (mg/dl)
carbohydrate metabolism | change from baseline insulin levels (UI/L) at 8 weeks
  change of seric carbohydrate parameters markers such as insulin levels (UI/L)
carbohydrate metabolism | change from baseline HOMA-Insulin Resistance (units) at 8 weeks
  change of seric carbohydrate parameters markers such as HOMA-Insulin resistance (units)
Blood pressure | change from baseline systolic blood pressure (mmHg) and diastolic blood pressure (mmHg) at 8 weeks
  change of systolic blood pressure (mmHg) and diastolic blood pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Daniel de Luis Roman, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No